CLINICAL TRIAL: NCT04237025
Title: Effects of Nordic Walking Exercise on Gait, Motor/Non-motor Symptoms, and Exercise Biomarkers in Individuals With Parkinson's Disease
Brief Title: Effects of Nordic Walking Exercise on Gait, Motor/Non-motor Symptoms, and Exercise Biomarkers in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Responsible Party: Principal Investigator, Cathy Harro, Associate Professor, Physical Therapy, Grand Valley State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-101-H
Record Dates: First submitted 2020-01-14; First posted 2020-01-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: exercise therapy; mobility limitation; walk test; biomarkers
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This study will employ a prospective, single cohort pre- and post-intervention research design. Supervised and individually prescribed Nordic Walking (NW) exercise will be conducted in a small group setting with a 2:1 participant to trainer ratio providing individualized instruction and progression of training. Training will be conducted for a total of 14 one-hour sessions over a 6-week period.
  In addition to the supervised NW training sessions, participants will be asked to complete independent NW exercise at least 2 times weekly during the 6-week training period. Following the completion of the 6-week supervised NW training period, participants will be asked to independently continue their NW exercise as least three times per week for the 3-month follow-up period. Independent NW exercise logs and adherence will be monitored during both the supervised training phase and the 3-month follow-up phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nordic walking exercise group (Experimental): Supervised Nordic walking exercise training 3 times per week for the first two weeks and 2 times per week for next four weeks (total 6 weeks). In addition to independent Nordic walking exercise twice weekly during intervention phase and three times weekly during the 3-month followup phase.
  Interventions: Other: Nordic walking exercise

INTERVENTIONS:
Other: Nordic walking exercise — Supervised Nordic Walking (NW) exercise will be conducted in a small group setting with a 2:1 participant to trainer ratio providing individualized training instruction. Training will be conducted for a total of 14 one-hour sessions over a 6-week period. Training will take place at an outdoor community track with progression tasks on hills or grassy terrain. The one-hour training sessions will include a 10-minute warm-up period, 45 minutes of individualized NW training, and a 5-minute cool down period. The target training duration goal for NW exercise will be 45 minutes of continuous walking at moderate intensity based on target heart rate and Rating of Perceived Exertion. NW exercise program will be customized and progressed for each participant by trainers with ongoing assessment of participant's gait pattern, NW technique, and exercise responses during the training sessions. Group comradery and accountability will be facilitated through training in small group training context.

SUMMARY:
The purpose of this study is to examine the effects of Nordic pole walking exercise on walking function, movement and non-movement Parkinson-related symptoms, and certain exercise-related chemical indicators (bio-markers) in people with Parkinson's disease.

This study will examine both the immediate and long-term effects of Nordic walking (NW) exercise on walking function, PD symptoms and exercise bio-markers after a supervised and individually progressed 6-week NW exercise training period and after a 3-month independent NW exercise phase.

NW, as a task- specific exercise with higher energy demands than regular walking, has good practicality for independent walking exercise once the training program is completed. Therefore, this study will also examine independent NW exercise engagement after a supervised training program to assess feasibility and sustainability of this mode of task-specific aerobic exercise.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a highly prevalent neuro-degenerative disorder in older adults that leads to reduced activity levels, physical disability, and accelerated age-related decline in mobility. Gait dysfunction and postural instability are key motor problems that develop with disease progression and adversely affect independent mobility, fall risk and activity participation. Prevention of balance, gait and functional decline are priority goals in physical therapy management for individuals with PD. Early activity-based and exercise interventions are supported as critical components for disease management and slowing disease progression. Furthermore, the underlying mechanisms by which exercise-based interventions effect changes in motor and non-motor symptoms in PD need to be further elucidated.

Individualized aerobic exercise prescription that is task-specific, challenging, and feasible for an independent exercise program is needed for individuals with PD to optimize their walking and motor function and sustain long-term engagement in regular physical exercise. Walking as a form of aerobic exercise has been reported to be safe in a community setting and to improve functional and gait outcomes and quality of life in PD. Nordic walking (NW) is a form of fitness walking using specialty poles that mimics the full body movement pattern of cross-country skiing, can be performed in varied terrains and may offer additional benefits beyond simple treadmill or over ground walking. NW technique has specific benefits for Parkinson gait, as it incorporates rhythmic timing of inter-limb coordination, increased engagement of upper extremities and upright trunk, and high energy expenditure resulting in a beneficial aerobic conditioning effect.

There is also consistent scientific evidence in both clinical and animal studies that shows the benefits of exercise at the cellular level in PD. Moderate to intense aerobic exercise enhances PD brain health and supports neural plasticity. Cellular changes include increased blood flow and angiogenesis, up-regulated neurotrophic factors, reduced neuro-inflammation, and enhanced immune responses. This project will evaluate the effects of NW in persons with PD at the molecular level with 3 known exercise-related bio-markers. These 3 bio-markers are brain-derived neurotropic factor (BDNF), cortisol, and alpha-amylase (α-amylase) proteins.

Study objectives:

Given the rapid accumulation of evidence showing the benefits of exercise in PD, there is a need to investigate which modes of exercise training have positive effects both on clinical measures and on bio-markers that are indicative of biochemical changes to support PD brain health. With a previously reported moderate aerobic conditioning effect following NW in both healthy elderly and PD cohorts, the premise is that this intensive fitness walking may produce changes at the cellular and molecular levels. Investigating changes in walking and motor/non-motor function following NW exercise and correlating these changes with exercise-related bio-markers may provide foundation support for the neuro-protective benefit of NW in persons with PD. Thus, the purpose of this proof-of concept study is to investigate the immediate and long-term effects of NW exercise on walking function, motor/non-motor PD symptoms and exercise-related bio-markers in persons with mild to moderate idiopathic PD. Additionally, this study will examine independent NW exercise engagement after a supervised training program to assess feasibility and sustainability of this mode of task-specific aerobic exercise.

Study Design:

This study will employ a prospective, single cohort pre- and post-intervention research design. Rationale for this design is twofold: 1. proof-of-concept in order to assess intervention effects based on functional and clinical measures following NW training and examine if these measures are associated with changes in exercise-related bio-markers in PD; and 2. assessment of feasibility of independent engagement in NW exercise after a supervised program in persons with mild to moderate PD as a mode of task-specific physical activity engagement. This research design will involve a 4-week baseline phase with two time points for assessment of dependent measures (T0-A and T0-B) to assess for a stable baseline, followed by a 6-week NW training intervention phase with a post-training assessment (T1) at the end of the 6 weeks, and a 3-month independent NW exercise phase with a follow-up assessment at the end of the 3 months (T2). Previous work in our lab has demonstrated significant improvements in walking and balance measures following a 6-week treadmill and rhythmic over ground auditory cuing protocols, and therefore, a 6-week training duration is expected to be sufficient for inducing training effects. Supervised NW adherence and independent NW exercise adherence, as well as any adverse effects will be monitored to determine feasibility and safety, particularly for independent NW phase of the study.

Data Analysis:

Descriptive statistics on patients' demographic characteristics (e.g. age, disease duration, stage, PD sub-type, fall history, activity level classification, medications and co-morbidity) will be documented. PD sub-type is categorized as tremor dominant, posture instability/gait difficulty, and indeterminate, based on MDS-UPDRS score. Descriptive statistics on patient's training sessions and training progression across the six weeks will be synthesized and analyzed. This training session data will include: training activities, walking speed, duration and distance of NW, Rating of Perceived Exertion, and walking terrain. Data from activity logs will be examined to reflect independent NW exercise adherence and activity level (number of steps/day) both during the 6-week training program and the follow-up independent exercise phase. Fall report data and any adverse events will be documented. This adherence and safety descriptive data during 3-month follow-up phase will reflect feasibility of independent home NW exercise program following a supervised NW training program.

Descriptive statistics for the gait, clinical PD-motor and non-motor, and bio-marker outcome measures will be calculated. Comparison of the two-baseline gait and clinical measures (Baseline-week 1 T0-A vs baseline week 4 T0-B) will be analyzed using dependent t-tests to determine if there was a stable baseline for these dependent measures. If analysis reveals no differences between baseline measures, then T0-B will be used for comparison to T1 and T2 measures. If analysis reveals differences between baseline measures, then the average of the two measures will be used for comparison to T1 and T2 measures. Dependent measures distribution across the three time points (T0, T1, T2) will be analyzed to assess if meet the assumption of normal distributions. If the data are normally distributed, one-way repeated measures analysis of variance (ANOVA) with planned contrasts will be used for each outcome measure to compare baseline to T1, baseline to T2, and T1 to T2. ANOVA is a statistical method to test differences between two or more means (mean = average of a data set). A repeated measures ANOVA can be used to determine whether there is any statistically significant difference between the means of three or related groups (in this study, a related group is a specific time point). IF normality assumptions are not met, then the Friedman test with post hoc Wilcoxon sign-ranked pairwise comparisons will be used for each outcome measure to compare baseline to T1, baseline to T2, and T1 to T2 timepoints. Bonferroni correction was applied due to the number of analyses being conducted. Level of significance was set at 0.05. Repeated measures ANOVA will also be used to assess the changes in means over 8 collection time points in the BDNF, cortisol, and α-amylase data and show a time-course of the NW exercise effects in persons with PD. P value was set at p <.05 for all statistical tests. To examine the magnitude of the training effects, the Cohen effect size will be calculated for those variables that demonstrated statistically significant change.

Raw data of gene expression will be normalized and background corrected to set the data set to a common scale and remove the effects of non-specific binding across the micro arrays. The Limma package in R, a computational programming language for statistical computing and graphics will be used. Differential-expressed genes can then be identified to show gene expression changes that are statistically significant between different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a diagnosis of idiopathic Parkinson disease
2. Parkinson medications and dosing must be unchanged over the past month
3. Must be residing in the community (eg... not supportive living or skilled nursing facility)
4. Must have the ability to safely and continuously ambulate a minimum distance of 500 feet independently without an assistive device
5. Must have the ability to ascend and descend a full flight of stairs with or without the use of railings with no more than stand by assistance
6. Must have functional vision with or without corrective lens for safe outdoor mobility

Exclusion Criteria:

1. Must have no other neurologic diagnoses (such as brain injury, multiple sclerosis or stroke)
2. Must have no significant comorbidities (cardiorespiratory conditions, orthopedic conditions, or recent orthopedic surgery) that would limit their ability to safely participate in an intensive walking exercise program
3. Must not have cognitive impairment as determined by a Montreal Cognitive Assessment score below 21 points
4. Must not have had recent deep brain stimulation (DBS) (within last 3 months) or planned DBS in next 4 months
5. Must not be previously trained in Nordic Walking technique And are currently engaged in moderate intensity Nordic Walking exercise at least 3 days per week

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
10 Meter Walk Test | Change from baseline gait speed at 6 weeks and at 3 months
  Comfortable and fast gait speed (m/s) conducted on measured level walkway using standardized procedures. 10-Meter walk test is the gold standard for assessment of the effectiveness of walking training interventions in PD
6-Minute Walk test | Change from baseline walking distance at 6 weeks and at 3 months
  Measures walking distance (m) using standardized 100 ft. walkway and procedures from American Thoracic Society. Measure reflects walking endurance and sub-maximal cardiovascular endurance. 6-Minute Walk test is a valid and reliable measure of walking function in persons with PD.
Temporal-distance gait measures | Change from baseline temporal gait measures at 6 weeks and at 3 months
  Computerized assessment of temporal gait measures: stride length, cadence, stride time variability. These gait measures are sensitive indicators of gait dysfunction in persons with Parkinson disease. This study will assess if Nordic walking exercise improves gait pattern and efficiency.
Timed Up and Go test (TUG) | Change from baseline TUG times at 6 weeks and at 3 months
  Timed Up & Go test and the Cognitive-TUG and Motor-TUG timed tests (seconds) are sensitive functional mobility and dual task measures in Parkinson disease. Dual task TUG measure has excellent specificity and sensitivity to identify fall risk in Parkinson disease.
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Change from baseline UPDRS score at 6 weeks and at 3 months
  The MDS-UPDRS is the gold standard for assessing disease severity in PD and is commonly used to measure treatment effectiveness. In this study the MDS-UPDRS will be used to assess motor and non-motor symptoms.
Revised-Freezing of Gait Questionnaire | Change from baseline score at 6 weeks and at 3 months.
  The revised Freezing of Gait Questionnaire will be administered to determine if participant is experiencing any freezing and if so, the frequency, severity and impact of freezing on their daily mobility. Minimum score=0; Maximum score=24; higher score reflects more severe freezing of gait.
Parkinson's Non-Motor Symptom Scale | Change from baseline score at 6 weeks and at 3 months.
  The Parkinson Non-Motor Symptom Scale is a self-report questionnaire used to assess the non-motor symptoms experienced by the individual during the past month. This is a valid measure of the effects of non-motor symptoms on daily function.Minimum score=0; Maximum score= 360; higher score is worse, reflects more symptoms.
Brain-derived neurotrophic factor (BDNF) | Change from baseline BDNF levels at 6 weeks and at 3 months.
  BDNF will be analyzed as a bio-marker to evaluate the potential neuro-protective effects of exercise in PD. Blood samples will be collected and both serum and plasma BDNF levels will be analyzed. Serum or plasma BDNF levels are currently used as proxy for BDNF central expression due to the difficulty to measure the levels in Central Nervous System.
Cortisol levels | Change from baseline Cortisol levels at 6 weeks and at 3 months.
  Cortisol levels are measured as exercise bio-markers. Cortisol levels may be reflective of stress and are related to neuro-inflammatory response in the nervous system. Saliva samples will be collected and analyzed for cortisol levels. Cortisol levels may be used as non-invasive stress-related bio-markers to gauge the effects of NW in persons with PD.
α-Amylase | Change from baseline α-Amylase levels at 6 weeks and at 3 months.
  α-Amylase will be analyzed as an exercise bio-marker. Reduced salivary α-amylase reflective of decreased stress reactivity has been reported after exercise intervention. α-Amylase are valuable non-invasive stress-related bio-markers to gauge the effects of NW in persons with PD.
Daily Physical Activity | Change (average daily steps) from baseline at 6 weeks and at 3 months followup.
  Average daily steps will be tracked by a Fitbit Inspire HR™ and documented. Average daily steps sampled from one week at baseline, at end of training phase (T-1) and followup phase (T-2).

SECONDARY OUTCOMES:
Parkinson's Fatigue Scale | Change from baseline score at 6 weeks and at 3 months. .
  Parkinson Fatigue Scale is a standardized questionnaire that assesses fatigue and its impact on daily function in individuals with PD. This tool will be used as secondary measure of any change in nonmotor symptoms following Nordic walking exercise. Minimum score=10; Maximum score=80; higher score is worse reflecting more severe fatigue symptoms
Percent Adherence to Independent Nordic Walking Exercise Sessions | At 3 months post-supervised Nordic Walking training
  Participants' completed Activity logs and use of activity monitors will be used to document and analyze exercise adherence (frequency, duration, intensity, and distance) of their NW weekly independent exercise and daily total number of steps. These measures will be reflective of NW adherence following supervised training period in the 3-month follow-up phase of the study.
Prospective Fall Report | At 3 months post-supervised Nordic walking training
  Participants will complete a monthly fall calendar to document any falls and near falls during the study duration. Prospective fall calendars are the gold standard for fall tracking and evidence shows that patients often forget and under-report falls when using a retrospective recall method. Fall report during the 3-month follow-up phase will be used to assess adverse events and safety of independent NW exercise in this sample.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy C Harro, DPT, MS, Principal Investigator — Grand Valley State University; Sok Kean Khoo, PhD, Principal Investigator — Grand Valley State University; Michael Shoemaker, DPT, PhD, Principal Investigator — Grand Valley State University
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
This proof of concept study is planned as a first step in examining effects of Nordic Walking on both functional and bio-marker outcomes; and will lay the foundation our next stage of research on this intervention.

REFERENCES:
- [Background] Ahlskog JE. Does vigorous exercise have a neuroprotective effect in Parkinson disease? Neurology. 2011 Jul 19;77(3):288-94. doi: 10.1212/WNL.0b013e318225ab66. PMID 21768599
- [Background] Flach A, Jaegers L, Krieger M, Bixler E, Kelly P, Weiss EP, Ahmad SO. Endurance exercise improves function in individuals with Parkinson's disease: A meta-analysis. Neurosci Lett. 2017 Oct 17;659:115-119. doi: 10.1016/j.neulet.2017.08.076. Epub 2017 Sep 1. PMID 28870627
- [Background] Ahlskog JE. Aerobic Exercise: Evidence for a Direct Brain Effect to Slow Parkinson Disease Progression. Mayo Clin Proc. 2018 Mar;93(3):360-372. doi: 10.1016/j.mayocp.2017.12.015. PMID 29502566
- [Background] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037
- [Background] Bombieri F, Schena F, Pellegrini B, Barone P, Tinazzi M, Erro R. Walking on four limbs: A systematic review of Nordic Walking in Parkinson disease. Parkinsonism Relat Disord. 2017 May;38:8-12. doi: 10.1016/j.parkreldis.2017.02.004. Epub 2017 Feb 6. PMID 28202374
- [Background] Cugusi L, Manca A, Dragone D, Deriu F, Solla P, Secci C, Monticone M, Mercuro G. Nordic Walking for the Management of People With Parkinson Disease: A Systematic Review. PM R. 2017 Nov;9(11):1157-1166. doi: 10.1016/j.pmrj.2017.06.021. Epub 2017 Jul 8. PMID 28694221
- [Background] Skorkowska-Telichowska K, Kropielnicka K, Bulinska K, Pilch U, Wozniewski M, Szuba A, Jasinski R. Nordic walking in the second half of life. Aging Clin Exp Res. 2016 Dec;28(6):1035-1046. doi: 10.1007/s40520-016-0531-8. Epub 2016 Jan 23. PMID 26803510
- [Background] Monteiro EP, Franzoni LT, Cubillos DM, de Oliveira Fagundes A, Carvalho AR, Oliveira HB, Pantoja PD, Schuch FB, Rieder CR, Martinez FG, Peyre-Tartaruga LA. Effects of Nordic walking training on functional parameters in Parkinson's disease: a randomized controlled clinical trial. Scand J Med Sci Sports. 2017 Mar;27(3):351-358. doi: 10.1111/sms.12652. Epub 2016 Feb 2. PMID 26833853
- [Background] Petzinger GM, Fisher BE, McEwen S, Beeler JA, Walsh JP, Jakowec MW. Exercise-enhanced neuroplasticity targeting motor and cognitive circuitry in Parkinson's disease. Lancet Neurol. 2013 Jul;12(7):716-26. doi: 10.1016/S1474-4422(13)70123-6. PMID 23769598
- [Background] Hirsch MA, van Wegen EEH, Newman MA, Heyn PC. Exercise-induced increase in brain-derived neurotrophic factor in human Parkinson's disease: a systematic review and meta-analysis. Transl Neurodegener. 2018 Mar 20;7:7. doi: 10.1186/s40035-018-0112-1. eCollection 2018. PMID 29568518
- [Background] Soares NM, Pereira GM, Altmann V, de Almeida RMM, Rieder CRM. Cortisol levels, motor, cognitive and behavioral symptoms in Parkinson's disease: a systematic review. J Neural Transm (Vienna). 2019 Mar;126(3):219-232. doi: 10.1007/s00702-018-1947-4. Epub 2018 Oct 29. PMID 30374595
- [Background] Smyth N, Skender E, David FJ, Munoz MJ, Fantuzzi G, Clow A, Goldman JG, Corcos DM. Endurance exercise reduces cortisol in Parkinson's disease with mild cognitive impairment. Mov Disord. 2019 Aug;34(8):1238-1239. doi: 10.1002/mds.27719. Epub 2019 May 20. No abstract available. PMID 31107979
- [Background] Masters JM, Noyce AJ, Warner TT, Giovannoni G, Proctor GB. Elevated salivary protein in Parkinson's disease and salivary DJ-1 as a potential marker of disease severity. Parkinsonism Relat Disord. 2015 Oct;21(10):1251-5. doi: 10.1016/j.parkreldis.2015.07.021. Epub 2015 Jul 23. PMID 26231472

DOCUMENTS (1):
  • Informed Consent Form (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT04237025/ICF_000.pdf